CLINICAL TRIAL: NCT06297707
Title: Effect of Aquatic High Intensity Resistive Training on Cardiac Function and Exercise Capacity in Patients With Chronic Heart Failure
Brief Title: Effect of Aquatic High Intensity Resistive Training on Patients With Chronic Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, marwa mahmoud elsayed mahmoud, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005044
Record Dates: First submitted 2024-02-22; First posted 2024-03-07 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): aquatic high intensity resistive training
  Interventions: Other: aquatic high intensity resistive training
- control group (Active Comparator): usual care
  Interventions: Other: usual care

INTERVENTIONS:
Other: aquatic high intensity resistive training — The experimental group participants will involve in aquatic high intensity resistive training sessions. The participants in the intervention group will receive 1 h of supervised lower limb aquatic resistance training three times a week for 12 weeks, for a total of 36 training sessions.
  Arms: experimental group
Other: usual care — The control group will maintain usual care and will be asked to continue their usual leisure time activities. They will be offered the possibility of participating in two sessions consisting of 1 h of light stretching and relaxation during the 3-month intervention period.
  Arms: control group

SUMMARY:
PURPOSE:

to evaluate effect of aquatic high intensity resistive training on cardiac function and exercise capacity in patients with chronic heart failure.

BACKGROUND:

Heart failure (HF) is a rapidly growing public health issue with an estimated prevalence of >37.7 million individuals globally. HF is a shared chronic phase of cardiac functional impairment secondary to many etiologies, and patients with HF experience numerous symptoms that affect their quality of life, including dyspnea, fatigue, poor exercise tolerance, and fluid retention.

DETAILED DESCRIPTION:
It is an interventional study in which 60 chronic heart failure patients estimated to enroll according to random allocation and divided into two groups. The experimental group participants will involve in aquatic high intensity resistive training sessions. The participants in the intervention group will receive 1 h of supervised lower limb aquatic resistance training three times a week for 12 weeks, for a total of 36 training sessions. Resistance of exercises will be progressed with three different levels: barefoot, small fins and large resistance boots and the training leg will perform all the movements without contact with the pool walls or bottom i.e., non-weight bearing. The intervention will be completed in small groups of 6-8 subjects in a pool heated to 30-32 with two instructors: one ensuring intensity and the other full range of movement. Intensity of the training sessions will be set at "as hard and fast as possible" to ensure maximal muscle contraction. Full range of motion will be strictly controlled for to ensure optimal movement of synovial fluid and exposure of the whole cartilage to the low compressive and shear forces created by the muscle contraction and movement. Training intensity will be monitored using heart rate monitors (Polar Electro Ltd, Kempele, Finland), rate of perceived exertion (RPE) using the Borg 6-20 scale and number of repetitions achieved per movement.

The control group will maintain usual care and will be asked to continue their usual leisure time activities. They will be offered the possibility of participating in two sessions consisting of 1 h of light stretching and relaxation during the 3-month intervention period.

ELIGIBILITY:
Inclusion Criteria:

Age ranges from 45 to 60 years old. Have chronic heart failure (NYHA class I to III).

* Left ventricular ejection fraction (LVEF) > 50%
* clinically stable with optimal pharmacological therapy in greater than three months
* All patients didn't participate in any rehabilitation programs prior to the study.

Exclusion Criteria:

Signs of acute heart failure, unstable angina, or severe arrhythmia three months prior to enrolment in the study.

Pacemakers. recently diagnosed acute coronary syndrome or a recent coronary intervention or both renal insufficiency (estimated glomerular filtration rate < 30 mL/min) liver abnormalities uncontrolled hypertension moderate-to-severe valvular disease uncompensated heart failure patients Chronic lung disease. Other disorders counteracting exercise conditions that limit lower limb mobility (for example, burns, fractures)

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Cardiac function | 12 weeks
  echocardiogram Left ventricular systolic dysfunction will be assessed using the ejection fraction by 2D simpson method (the percentage of the end diastolic volume ejected during systole

SECONDARY OUTCOMES:
exercise capacity | 12 weeks
  6 minute walk test distance
physical symptoms of heart failure | 12 weeks
  Minnesota Living with Heart Failure Questionnaire The questionnaire has 21 items. Assessing the impact of frequent physical symptoms of heart failure

CONTACTS AND LOCATIONS:
Overall Officials: marwa elsayed, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy, Cairo, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Yes
sharing study protocol with other researches
Supporting Information: Study Protocol
Time Frame: 2 years
Access Criteria: acceptance the publishing journal
URL: http://www.ekb.com